CLINICAL TRIAL: NCT07263061
Title: Time to Post-operative Recovery of Serum Albumin as a Predictor of Outcome in Major Hepato Pancreato Biliary Surgeries
Status: Recruiting | Type: Observational
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Other Study IDs: IEC/2024/110/MA04
Record Dates: First submitted 2025-11-22; First posted 2025-12-04 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-11

CONDITIONS: Hepatobiliary Disease; Pancreas Disease; Bile Duct Diseases
MeSH Terms: conditions — Digestive System Diseases; Pancreatic Diseases; Bile Duct Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- hepatobiliary and pancreatic diseases: Patients undergoing Major Hepato Pancreato biliary surgeries
  Interventions: Other: NO TREATMENT

INTERVENTIONS:
Other: NO TREATMENT — NO TREATMENT

SUMMARY:
Hepatobiliary and Pancreatic surgery is associated with substantial risk of postoperative complications. Albumin is a negative acute phase protein. Its rapid decline may be due to degree of inflammation due to surgical procedures. The decline may due to multifactorial causes. Currently, contemporary data regarding the time to recovery of albumin, as a marker for early recovery of patient from surgical stress is sparse. Delta albumin is influenced by perioperative fluid administration and albumin supplementation. Delta albumin may not reflect the true surgical stress. Early post op albumin is a reflection of intraoperative events and not postoperative recovery or events and is unpredictable. Shorter recovery time of albumin is associated with less post op complications and hospital stay. Earlier recovery of albumin predicts lower morbidity and shorter hospital stay.

DETAILED DESCRIPTION:
Hepatobiliary and Pancreatic surgery is associated with substantial risk of postoperative complications. Albumin is a negative acute phase protein. Its rapid decline may be due to degree of inflammation due to surgical procedures. The decline may due to multifactorial causes. Currently, contemporary data regarding the time to recovery of albumin, as a marker for early recovery of patient from surgical stress is sparse. Delta albumin is influenced by perioperative fluid administration and albumin supplementation. Delta albumin may not reflect the true surgical stress.

ELIGIBILITY:
Inclusion Criteria:

1. All patients undergoing major Hepato pancreatico Biliary surgeries.
2. Patients who are more than 12 years of age
3. Retrospective arm - Data from 2010

Exclusion Criteria:

1. Patients who refuse or are unable to give consent.
2. Patients with Nephrotic syndrome, Protein losing enteropathies, Inflammatory bowel
3. Disease, Chronic Liver Disease.
4. Emergency Surgeries

Ages: 13 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients undergoing major Hepato pancreatico Biliary surgeries.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-12-07 (Actual); Primary Completion 2026-10-23 (Estimated); Study Completion 2026-10-23 (Estimated)

PRIMARY OUTCOMES:
Time to recovery of serum albumin as a predictor of outcome in major hepatobiliary surgeries as measured by hospital stay. | 30 days
  Time taken for unsupported albumin in Liver function test in a rising trend (g/dl)

SECONDARY OUTCOMES:
To correlate the time to recovery of albumin with complications and morbidity (Clavien Dindo classification, Comprehensive Complication Index, Intensive Care Unit Stay) | 30 days
  Major Complications measured by Clavien Dindo Classification (Major >grade 3A) and Comprehensive complication index (Major More than 27)
Time to reversal trend of albumin and Hospital stay | 30 days
  Time taken for unsupported albumin in Liver function test to reach a value of more than 3 g/dl and compared with the hospital stay
correlation of time to recovery of albumin and re admission rates | 90 days
  Time taken for unsupported albumin in Liver function test to reach a value of more than 3 g/dl and compared with the 90 day re admission rates

CONTACTS AND LOCATIONS:
Overall Officials: Dr Ragini Kilambi, MCh, Study Director — ILBS
Locations (1):
- ILBS, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided